CLINICAL TRIAL: NCT00431314
Title: The Effect of Hemodialysis on Toe Pressure- and Finger Pressure Measurements and Measurement of Skin Autofluorescence; a Pilot Study in the Assessment of Critical Limb Ischemia in Hemodialysis Patients.
Brief Title: Effect of Hemodialysis on Toe Pressure- and Finger Pressure and Skin Autofluorescence in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Isala (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Dutch research foundation
Other Study IDs: HD
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2007-01

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease; Hemodialysis; Critical Limb Ischemia; Autofluorescence
MeSH Terms: conditions — Kidney Failure, Chronic; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine the vascular condition of hemodialysis patients with toe pressure measurement, finger pressure measurement and measuring glycated and oxidated proteins by skin autofluorescence.

Hypothesis: Lowering of finger pressure/toe pressure during hemodialysis, especially in whom with a arteriovenous fistula, may contribute to critical limb ischemia in the extremities.

DETAILED DESCRIPTION:
1. To determine the macrovascular status of hemodialysis patients by measuring toe pressure, finger pressure and skin autofluorescence.
2. Measuring toe- and finger pressure before and during hemodialysis to determine the chance of developing critical limb ischemia in the extremities.
3. To assess the differences in finger pressure in hemodialysis patients before and during hemodialysis in patients with either arteriovenous fistula in the upper extremity or not.
4. To predict mortality and cardiovascular disease by determine the fastness of accumulation of Advanced-Glycation-Endproducts (this concerns follow-up measurements of skin autofluorescence; another study has collected data of skin autofluorescence in hemodialysis patients in our centre in 2003)

ELIGIBILITY:
Inclusion Criteria:

* Patients with End Stage Renal Disease with hemodialysis therapy

Exclusion Criteria:

* Hemodialysis during the night
* Dark coloured skin towards unreliable skin autofluorescence measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis patients in one hemodialysis centre
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2007-01; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henk J Bilo, PhD, Study Director — Center of Excellence Diabetes